CLINICAL TRIAL: NCT04989361
Title: Clinical Controlled Study and Safety Evaluation of the Therapeutic Effect of Soluble Hyaluronic Acid Microneedle and Non-ablative Fractional Laser on Infraorbital Wrinkles
Brief Title: Soluble Hyaluronic Acid Microneedle VS. Non-ablative Fractional Laser on Infraorbital Wrinkles.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Professer, Shanghai Dermatology Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiDH
Record Dates: First submitted 2021-06-18; First posted 2021-08-04 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Wrinkle
Keywords: microneedle; non-ablative fractional laser

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedle side (Experimental): Apply soluble hyaluronic acid microneedle eye mask to the periorbital area after normal facial cleansing and skin care every night for 20 days. Press and hold for 3 minutes, and then remove it after 1 h. Every 2 days for the next 20 days, and every 3 days for the last 21 days. Follow-up time: every 20 days during the treatment period, and follow-up visits in the 2nd, 4th, 8th and 12th weeks after the treatment.
  Interventions: Procedure: Soluble Hyaluronic Acid Microneedle
- Non-fractional laser side (Active Comparator): The patient received non-ablative fractional laser treatment once. Follow-up time: follow-up visits in the 2nd, 4th, 8th and 12th weeks after the treatment.
  Interventions: Procedure: Non-fractional laser

INTERVENTIONS:
Procedure: Soluble Hyaluronic Acid Microneedle — The soluble hyaluronic acid microneedle eye mask is a nanometer-sized microneedle made of water-soluble hyaluronic acid, which can directly inject the active ingredients into the dermis, and after being absorbed and dissolved by the skin, it can achieve the purpose of improving the water content and elasticity of the skin.
  Arms: Microneedle side
Procedure: Non-fractional laser — he non-ablative fractional laser use 1565nm fiber laser, which acts on the target base in the dermis-water. The beam penetrates the epidermis and acts on the dermis. Using the principle of focal light and heat, the tissue cells are heated to initiate the repair process, which promotes increased collagen synthesis, thereby Achieve the effect of firming the skin and improving wrinkles.
  Arms: Non-fractional laser side

SUMMARY:
This study is a prospective half-face controlled study, aiming to evaluate the therapeutic effects and adverse reactions of soluble hyaluronic acid microneedle and non-ablative fractional laser on infraorbital wrinkles and compare them.

DETAILED DESCRIPTION:
This study is a prospective half-face controlled study, aiming to evaluate the therapeutic effects and adverse reactions of soluble hyaluronic acid microneedle and non-ablative fractional laser on infraorbital wrinkles and compare them. The therapy is as follows:

1. Sign the informed consent form, and then the researchers will include and exclude patients according to the standards;
2. The researcher will collect the medical history, evaluate the condition, and determine the treatment plan after grouping by the random table;
3. Basic information collection 1) Take VISIA images (3 pictures of the front and sides at 45 degrees and several pictures of the skin lesions), and number and record the feature counts and specific scores of bilateral orbital wrinkles; 2) Measure and record the water content of the patient's periorbital skin;
4. Half face controlled treatment:

1) Drug preparation Drug: soluble hyaluronic acid microneedles; Equipment: ResurFX; 2) Treatment methods and operating procedures Microneedle side: Apply soluble hyaluronic acid microneedle eye mask to the periorbital area after normal facial cleansing and skin care every night for 20 days . Press and hold for 3 minutes, and then remove it after 1 h. Every 2 days for the next 20 days, and every 3 days for the last 21 days. Follow-up time: every 20 days during the treatment period, and follow-up in the second, fourth, eighth and twelfth week after the treatment.

Non-fractional laser side: The patient received non-ablative fractional laser treatment once. Follow-up time: follow-up visits in the 2nd, 4th, 8th and 12th weeks after the treatment.

3) End point of treatment Microneedle side: The soluble hyaluronic acid microcrystalline eye mask was used for 61 days according to the prescribed protocol. After the treatment, the patient entered the follow-up.

Fractional laser side: After one treatment, the patient enters the follow-up.

5. Follow-up after treatment Follow-up time: 2 weeks, 4 weeks, 8 weeks, 12 weeks after the end of treatment; Follow-up content: According to the follow-up plan, it is recommended that patients actively come to the hospital for follow-up. The follow-up time starts from the first day after the end of the last treatment. Record the patient's name, gender, age, adverse reactions, etc. in detail, take VISIA photos; test and record the skin moisture content, and fill in the patient satisfaction survey in the 4th week after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old, Skin Aging Atlas: Volume 2, Asian type infraorbital wrinkles assessment standard score 3 points and above;
2. After fully explaining the purpose and content of this clinical trial (including the subjects' compliance, etc.), on the basis of full understanding, voluntarily sign an informed consent to participate in the clinical trial.

Exclusion Criteria:

1. Those who are known to be allergic to test drugs or related drugs;
2. Pregnant or lactating women;
3. Received wrinkle treatment (laser, radio frequency, fruit acid, photon, hyaluronic acid filling, etc.) within 6 months before enrollment;
4. Those who have other diseases (infection, dermatitis, sunburn, scars, etc.) that may affect the evaluation of the efficacy of the facial treatment area and nearby areas;
5. Received anti-inflammatory, glucocorticoid or tretinoin treatment within 1 month before enrollment;
6. Participate in any drug clinical trial (as a subject) within 1 month before participating in this trial;
7. Combined with serious diseases, including severe heart disease,cerebrovascular disease, uncontrolled diabetes, uncontrolled high blood pressure, etc.;
8. Those with scar constitution;
9. Subjects with severe physical or mental illness that the investigator believes may affect treatment, evaluation, or poor compliance with the research protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Effective rate | 4 weeks after the treatment
  The grade of infraorbital wrinkles is assessed by a visual scale. Effective rate is defined as the proportion of patients who get improvement of at least one grade.

SECONDARY OUTCOMES:
Adverse reaction rate | Within 12 weeks after the treatment
  The adverse reaction is recorded during the study, including erythema, edema, crust, inch and pain. Adverse reaction rate is defined as the proportion of patients who have these reactions respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No